CLINICAL TRIAL: NCT03549767
Title: Randomized Trial to Compare Magnesium Sulphate Administration for Preeclampsia and Eclampsia: Springfusor Versus Standard of Approach
Brief Title: Springfusor for Administration of Magnesium Sulphate in Preeclampsia and Eclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 2018-015
Record Dates: First submitted 2018-02-27; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Preeclampsia and Eclampsia
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study is testing the acceptability of the device (springfusor) in the administration of magnesium suphate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Springfusor (Experimental): Women in this group will have their loading dose (4 gm of 50% Magnesium sulphate in 10 ml syringe administered over 20 minutes) and maintenance therapy (4 gm of 50% Magnesium sulphate in 10 ml syringe administered over 4 hours through an IV infusion administered using a Springfusor pump.. The 4 gm maintenance dose will be repeated every 4 hours for 24 hours.
  Interventions: Device: Springfusor
- Standard of care (Active Comparator): The control group will have Magnesium sulphate administered using the Pritchard regimen, which involves administration of loading dose of 4 gm of 20% Magnesium sulphate IV over 15-20 minutes, immediately followed by 10 gm of 50% Magnesium sulphate IM (5gm on each buttock). The maintenance dose of 5 gm of 50% Magnesium sulphate IM every 4 hourly in alternate buttocks continued for 24 hours
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Device: Springfusor — Springfusor for administration of magnesium sulphate
  Arms: Springfusor
Procedure: Standard of care — Pritchard regimen. Magnesium sulphate is administered using hospital practice
  Arms: Standard of care

SUMMARY:
Magnesium Sulphate is the drug of choice for prevention and treatment of seizures in preeclampsia and eclampsia. It is administered parenterally by intravenous (IV) and or intramuscular (IM) routes. The IM regimen requires repeated painful injections which may be a barrier to optimal utilization whereby, there is frequent omission of some doses or increased interval between maintenance doses and low patient acceptability of magnesium. The study plans to assess the acceptability and safety of Springfusor device in the administration of magnesium sulphate in preeclampsia and eclampsia.

DETAILED DESCRIPTION:
The IM regimen used in low resource settings, requires repeated painful injections which may be a barrier to optimal utilization whereby, there is frequent omission of some doses or increased interval between maintenance doses and low patient acceptability of magnesium. The study plans to assess the acceptability and safety of Springfusor device in the administration of magnesium sulphate in preeclampsia and eclampsia.

It is open label clinical randomized trail conducted at Mulago national referral and teaching hospital, where, 482 women diagnosed with preeclampsia and eclampsia will be randomized in blocks to either Springfusor device or standard of care for the administration of magnesium sulphate.

Women in the Springfusor group will have their loading dose (4 gm of 50% Magnesium sulphate in 10 ml syringe administered over 20 minutes) and maintenance therapy (4 gm of 50% Magnesium sulphate in 10 ml syringe administered over 4 hours. The 4 gm maintenance dose will be repeated every 4 hours for 24 hours) of Magnesium sulphate through an IV infusion administered using a Springfusor pump.

The control group will have Magnesium sulphate administered according to the Pritchard regimen (standard hospital practice). The Pritchard regimen involves administration of loading dose of 4 gm of 20% Magnesium sulphate IV over 15-20 minutes, immediately followed by 10 gm of 50% Magnesium sulphate IM (5gm on each buttock). The maintenance dose of 5 gm of 50% Magnesium sulphate IM every 4 hourly in alternate buttocks continued for 24 hours.

The primary outcome is the acceptability of administration of Magnesium sulphate using Springfusor assessed using a Likert scale. The other outcomes are discontinuation and complications in the two arms. Analysis will be intention to treat.

ELIGIBILITY:
Inclusion Criteria:

1. The study will include pregnant women with age of 15 years and above
2. Pregnancy of 20+ weeks of gestation or delivered within 24 hours,
3. Presenting with preeclampsia and eclampsia i.e. have a raised blood pressure (systolic of >140 mmHg and diastolic > 90mmHg), proteinuria >1+.
4. Presenting within the study period
5. Consent to participate in the study.

Exclusion Criteria:

1. Pregnant women or delivered within 24 hours who admitted with had received magnesium sulphate 24 hours prior to admission,
2. Has known allergy to magnesium sulphate and
3. Has elevated serum creatinine (>1.2 mg/dl). However the participants may be enrolled prior to the knowledge of serum creatinine, but withdrawn if the level is >1.2 mg/dl.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Springfusor | At 24 hours after loading dose
  Acceptability of Springfusor for administration of magnesium sulphate will be assessed using a Likert scale ranging from one (very acceptable) to five (very unacceptable).

SECONDARY OUTCOMES:
Discontinuation | 24 hour after the loading dose
  assessed as study participants who do not completed doses of magnesium sulphate
Level of pain | At 24 hours after loading dose
  The study participants will be asked to assess the severity of pain during the administration of magnesium sulphate using Visual analogue scale 1-7.
Safety of springfusor | within 24 hours
  Occurrence of respiratory depression eg rate <16/min

CONTACTS AND LOCATIONS:
Overall Officials: Sam Ononge, PhD, Principal Investigator — Makerere University College of Health Sciences
Locations (1):
- Mualgo Hospital, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037